CLINICAL TRIAL: NCT04942236
Title: Collaborative Model of Care Between Orthopaedics and Allied Health Care Professionals (CONNACT) OA Knee Cohort
Brief Title: CONNACT OA Knee Cohort
Acronym: CONNACT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: National Healthcare Group, Singapore (Other Government); Khoo Teck Puat Hospital (Other); Woodlands Health Campus (Other Government)
Responsible Party: Principal Investigator, Bryan Tan, Associate Consultant, Tan Tock Seng Hospital
Other Study IDs: WHC/2020-00076
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CONNACT OA knee cohort is a prospective longitudinal cohort study where we aim to collect sociodemographic, psychosocial, clinical, health utilization and cost data in order to better understand the Asian OA knee cohort and investigate for prognostic variables that can potentially influence a patients clinical outcome and treatment decisions.

In addition, the CONNACT OA knee cohort will form the basis for a cohort multiple randomized control trial (cmRCT) study design where multiple interventions can be tested in a randomized fashion. Each intervention is offered to a randomly selected sample of patients eligible for that intervention, who are then compared with the rest of the eligible patients from the cohort that are still being treated as usual.

ELIGIBILITY:
Inclusion Criteria:

1. Knee Osteoarthritis (based on NICE guidelines)
2. Age > 45 years
3. Community ambulator with or without walking aid
4. Conversant in English or Chinese

Exclusion Criteria:

1. Alternative diagnosis to Knee OA e.g. referred pain from spine or hip
2. Other forms of knee arthritis e.g. inflammatory, post-traumatic
3. Moderate to severe cognitive impairment e.g. dementia
4. Previous knee arthroplasty
5. Wheelchair bound patients
6. Medical conditions that will medically interfere with rehabilitation involvement e.g. decompensated heart failure, stroke with significant deficit, end stage renal failure

Ages: 46 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee Osteoarthritis patients for conservative treatment
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS-12) | Baseline
  Derived from the original 42-item Knee injury and Osteoarthritis Outcome Score (KOOS), KOOS-12 reduces respondent burden by 70% from the original KOOS while providing scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. The KOOS sub scales are scored using the method of summated ratings and transformed to range from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problem. The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. It also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.
Knee Injury and Osteoarthritis Outcomes Score (KOOS-12) | Change from Baseline to 3 months
  Derived from the original 42-item Knee injury and Osteoarthritis Outcome Score (KOOS), KOOS-12 reduces respondent burden by 70% from the original KOOS while providing scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. The KOOS sub scales are scored using the method of summated ratings and transformed to range from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problem. The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. It also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.
Knee Injury and Osteoarthritis Outcomes Score (KOOS-12) | Change from Baseline to 6 months
  Derived from the original 42-item Knee injury and Osteoarthritis Outcome Score (KOOS), KOOS-12 reduces respondent burden by 70% from the original KOOS while providing scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. The KOOS sub scales are scored using the method of summated ratings and transformed to range from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problem. The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. It also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.
Knee Injury and Osteoarthritis Outcomes Score (KOOS-12) | Change from Baseline to 12 months
  Derived from the original 42-item Knee injury and Osteoarthritis Outcome Score (KOOS), KOOS-12 reduces respondent burden by 70% from the original KOOS while providing scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact. The KOOS sub scales are scored using the method of summated ratings and transformed to range from 0 to 100, with 0 representing extreme knee problems and 100 representing no knee problem. The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. It also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Function, QoL | Baseline
  The three subscales of KOOS-12 are scored separately: KOOS Pain (4 items); KOOS Function (4 items); KOOS QoL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the three scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Function, QoL | Change from Baseline to 3 months
  The three subscales of KOOS-12 are scored separately: KOOS Pain (4 items); KOOS Function (4 items); KOOS QoL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the three scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Function, QoL | Change from Baseline to 6 months
  The three subscales of KOOS-12 are scored separately: KOOS Pain (4 items); KOOS Function (4 items); KOOS QoL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the three scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
Knee Injury and Osteoarthritis Outcomes Score (KOOS) subscales - Pain, Function, QoL | Change from Baseline to 12 months
  The three subscales of KOOS-12 are scored separately: KOOS Pain (4 items); KOOS Function (4 items); KOOS QoL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the three scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
EuroQol-5 Dimensions (EQ-5D) | Baseline
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
EuroQol-5 Dimensions (EQ-5D) | Change from Baseline to 3 months
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
EuroQol-5 Dimensions (EQ-5D) | Change from Baseline to 6 months
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
EuroQol-5 Dimensions (EQ-5D) | Change from Baseline to 12 months
  EuroQol-5 Dimensions (EQ-5D) consists of 2 dimensions, the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by selecting the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS will be used as a quantitative measure of health outcome.
Patient Health Questionnaire 4 (PHQ-4) | Baseline
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all', 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggest anxiety. Total score ≥3 for last 2 questions suggest depression.
Patient Health Questionnaire 4 (PHQ-4) | Change from Baseline to 3 months
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all', 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggest anxiety. Total score ≥3 for last 2 questions suggest depression.
Patient Health Questionnaire 4 (PHQ-4) | Change from Baseline to 6 months
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all', 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggest anxiety. Total score ≥3 for last 2 questions suggest depression.
Patient Health Questionnaire 4 (PHQ-4) | Change from Baseline to 12 months
  Measurement for depression and anxiety rated on a 4 point Likert-type scale. 0 refers to 'Not at all', 3 refers 'Nearly everyday'. Total score is determined by adding together the scores of each of the 4 items. Scores are rated as normal (0-2), mild (3-5), moderate (6-8), and severe (9-12).
  Total score ≥3 for first 2 questions suggest anxiety. Total score ≥3 for last 2 questions suggest depression.
Pain, Enjoyment, General Activity Scale (PEG) | Baseline
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain', 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.
Pain, Enjoyment, General Activity Scale (PEG) | Change from Baseline to 3 months
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain', 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.
Pain, Enjoyment, General Activity Scale (PEG) | Change from Baseline to 6 months
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain', 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.
Pain, Enjoyment, General Activity Scale (PEG) | Change from Baseline to 12 months
  Measures the pain intensity and interference level using a three-item scale. Scale of 0 to 10 is used for each item. 0 refers 'no pain', 10 refers 'worse pain'. Add the responses to the three questions, then divide by three to get a mean score (out of 10) on overall impact of points.

OTHER OUTCOMES:
OsteoArthritis Quality Indicator (OA QI) | Baseline
  The 17-items OA-QI questionnaire includes quality indicators related to patient education and information, assessment of pain and function, referrals, and pharmacologic treatment for OA. This questionnaire is administer at patient's baseline visit, after consultation with an orthopaedic surgeon, to find out patient-perceived quality of OA management. Using this outcome to investigate the quality of care delivered in primary and secondary care for patients with knee OA.
University of California, Los Angeles (UCLA) activity score | Baseline
  1 question survey to understands patient physical activity level from a scale of 1 (wholly inactive) to 10 (regular participation in impact sports).
University of California, Los Angeles (UCLA) activity score | Change from Baseline to 3 months
  1 question survey to understands patient physical activity level from a scale of 1 (wholly inactive) to 10 (regular participation in impact sports).
University of California, Los Angeles (UCLA) activity score | Change from Baseline to 6 months
  1 question survey to understands patient physical activity level from a scale of 1 (wholly inactive) to 10 (regular participation in impact sports).
University of California, Los Angeles (UCLA) activity score | Change from Baseline to 12 months
  1 question survey to understands patient physical activity level from a scale of 1 (wholly inactive) to 10 (regular participation in impact sports).
Global perceived effect (GPE) | 3 months
  Patient will be asked to rate thier overall recovery on a 7-point Likert scale. 1 refers to 'Very much improved'; 7 refers to 'Very much deteriorated'.
Global perceived effect (GPE) | 6 months
  Patient will be asked to rate thier overall recovery on a 7-point Likert scale. 1 refers to 'Very much improved'; 7 refers to 'Very much deteriorated'.
Global perceived effect (GPE) | 12 months
  Patient will be asked to rate thier overall recovery on a 7-point Likert scale. 1 refers to 'Very much improved'; 7 refers to 'Very much deteriorated'.
Patient Acceptable Symptom State (PASS) | 3 months
  A single-question used to assess patient's satisfaction in the treatment. Response will be either yes or no. "When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life."
Patient Acceptable Symptom State (PASS) | 6 months
  A single-question used to assess patient's satisfaction in the treatment. Response will be either yes or no. "When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life."
Patient Acceptable Symptom State (PASS) | 12 months
  A single-question used to assess patient's satisfaction in the treatment. Response will be either yes or no. "When you think of your knee function, will you consider your current condition as satisfying? By knee function, you should take into account your activities of daily living, sport and recreational activities, your pain and other symptoms and your quality of life."
Self-reported treatment failure | 3 months
  Patient who answers 'no' to PASS will be asked to determine if they consider the treatment to have failed. Response will be 'yes' or 'no'. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?"
Self-reported treatment failure | 6 months
  Patient who answers 'no' to PASS will be asked to determine if they consider the treatment to have failed. Response will be 'yes' or 'no'. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?"
Self-reported treatment failure | 12 months
  Patient who answers 'no' to PASS will be asked to determine if they consider the treatment to have failed. Response will be 'yes' or 'no'. "Would you consider your current state as being so unsatisfactory that you consider the treatment to have failed?"
Cumulative Analgesia Consumption Score (CACS) | 3 months
  Objective measurement of patient's analgesics average weekly consumption based on the quantity multiplied by the category of analgesic medication according to the WHO pain relief ladder (1 point - non-opioid, 2 points - mild opioid, 3 points - strong opioid) in order to calculate a total score.
Cumulative Analgesia Consumption Score (CACS) | 6 months
  Objective measurement of patient's analgesics average weekly consumption based on the quantity multiplied by the category of analgesic medication according to the WHO pain relief ladder (1 point - non-opioid, 2 points - mild opioid, 3 points - strong opioid) in order to calculate a total score.
Cumulative Analgesia Consumption Score (CACS) | 12 months
  Objective measurement of patient's analgesics average weekly consumption based on the quantity multiplied by the category of analgesic medication according to the WHO pain relief ladder (1 point - non-opioid, 2 points - mild opioid, 3 points - strong opioid) in order to calculate a total score.
Short dietary questionnaire | Baseline
  This questionnaire is to assess the eating habits and dietary choices over a period of time. It consists of 9 questions looking at the frequency of consumption in these categories - sugar, fats, fruits and vegetables, and wholegrains - and the degree of mindfulness in eating.
Short dietary questionnaire | Change from Baseline to 3 months
  This questionnaire is to assess the eating habits and dietary choices over a period of time. It consists of 9 questions looking at the frequency of consumption in these categories - sugar, fats, fruits and vegetables, and wholegrains - and the degree of mindfulness in eating.
Short dietary questionnaire | Change from Baseline to 6 months
  This questionnaire is to assess the eating habits and dietary choices over a period of time. It consists of 9 questions looking at the frequency of consumption in these categories - sugar, fats, fruits and vegetables, and wholegrains - and the degree of mindfulness in eating.
Short dietary questionnaire | Change from Baseline to 12 months
  This questionnaire is to assess the eating habits and dietary choices over a period of time. It consists of 9 questions looking at the frequency of consumption in these categories - sugar, fats, fruits and vegetables, and wholegrains - and the degree of mindfulness in eating.
Questionnaire measuring the direct and indirect costs | 3 months
  Cost questionnaire
Questionnaire measuring the direct and indirect costs | 6 months
  Cost questionnaire
Questionnaire measuring the direct and indirect costs | 12 months
  Cost questionnaire
Arthritis Self-efficacy scale 8 (ASES-8) | Baseline
  This 8-items shortened version of the original 20-item instrument includes two items from the pain subscale, four items from the other symptoms subscale, and two new items that relate to preventing pain and fatigue from interfering with daily activities. The questionnaire measures patients' confidence on a scale of 1 (very uncertain) to 10 (very certain) in their ability to manage symptoms of arthritis. Responses were averaged to yield a score ranging from 1 to 10, the higher number being having greater self-efficacy.
Arthritis Self-efficacy scale 8 (ASES-8) | Change from Baseline to 3 months
  This 8-items shortened version of the original 20-item instrument includes two items from the pain subscale, four items from the other symptoms subscale, and two new items that relate to preventing pain and fatigue from interfering with daily activities. The questionnaire measures patients' confidence on a scale of 1 (very uncertain) to 10 (very certain) in their ability to manage symptoms of arthritis. Responses were averaged to yield a score ranging from 1 to 10, the higher number being having greater self-efficacy.
Arthritis Self-efficacy scale 8 (ASES-8) | Change from Baseline to 6 months
  This 8-items shortened version of the original 20-item instrument includes two items from the pain subscale, four items from the other symptoms subscale, and two new items that relate to preventing pain and fatigue from interfering with daily activities. The questionnaire measures patients' confidence on a scale of 1 (very uncertain) to 10 (very certain) in their ability to manage symptoms of arthritis. Responses were averaged to yield a score ranging from 1 to 10, the higher number being having greater self-efficacy.
Arthritis Self-efficacy scale 8 (ASES-8) | Change from Baseline to 12 months
  This 8-items shortened version of the original 20-item instrument includes two items from the pain subscale, four items from the other symptoms subscale, and two new items that relate to preventing pain and fatigue from interfering with daily activities. The questionnaire measures patients' confidence on a scale of 1 (very uncertain) to 10 (very certain) in their ability to manage symptoms of arthritis. Responses were averaged to yield a score ranging from 1 to 10, the higher number being having greater self-efficacy.
Brief Fear of Movement Scale for Osteoarthritis | Baseline
  This scale will be used to assess fear of pain. It is based on the widely used Tampa Scale of Kinesiophobia and contains 6 questions that evaluate fear of pain, movement and re-injury. The patient is asked to indicate 1 (strongly disagree), 2 (disagree), 3 (agree) or 4 (strongly agree) for each item. The higher number represents increasing fear.
Brief Fear of Movement Scale for Osteoarthritis | Change from Baseline to 3 months
  This scale will be used to assess fear of pain. It is based on the widely used Tampa Scale of Kinesiophobia and contains 6 questions that evaluate fear of pain, movement and re-injury. The patient is asked to indicate 1 (strongly disagree), 2 (disagree), 3 (agree) or 4 (strongly agree) for each item. The higher number represents increasing fear.
Brief Fear of Movement Scale for Osteoarthritis | Change from Baseline to 6 months
  This scale will be used to assess fear of pain. It is based on the widely used Tampa Scale of Kinesiophobia and contains 6 questions that evaluate fear of pain, movement and re-injury. The patient is asked to indicate 1 (strongly disagree), 2 (disagree), 3 (agree) or 4 (strongly agree) for each item. The higher number represents increasing fear.
Brief Fear of Movement Scale for Osteoarthritis | Change from Baseline to 12 months
  This scale will be used to assess fear of pain. It is based on the widely used Tampa Scale of Kinesiophobia and contains 6 questions that evaluate fear of pain, movement and re-injury. The patient is asked to indicate 1 (strongly disagree), 2 (disagree), 3 (agree) or 4 (strongly agree) for each item. The higher number represents increasing fear.
Chronic illness-related shame score (CISS) | Baseline
  This 7-items shame score aim to find out the participants' shame feelings derived from chronic illness-related experiences. Each item is rated on a 5-point Likert (0: Never True; 4: Always True). Higher scores reveal higher levels of shame specifically associated with the experience of having an illness and/or its symptomatology.
Chronic illness-related shame score (CISS) | Change from Baseline to 3 months
  This 7-items shame score aim to find out the participants' shame feelings derived from chronic illness-related experiences. Each item is rated on a 5-point Likert (0: Never True; 4: Always True). Higher scores reveal higher levels of shame specifically associated with the experience of having an illness and/or its symptomatology.
Chronic illness-related shame score (CISS) | Change from Baseline to 6 months
  This 7-items shame score aim to find out the participants' shame feelings derived from chronic illness-related experiences. Each item is rated on a 5-point Likert (0: Never True; 4: Always True). Higher scores reveal higher levels of shame specifically associated with the experience of having an illness and/or its symptomatology.
Chronic illness-related shame score (CISS) | Change from Baseline to 12 months
  This 7-items shame score aim to find out the participants' shame feelings derived from chronic illness-related experiences. Each item is rated on a 5-point Likert (0: Never True; 4: Always True). Higher scores reveal higher levels of shame specifically associated with the experience of having an illness and/or its symptomatology.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline
  This scale is a 12-item questionnaire to identify the patients' perceived adequacy of social support from three sources: family, friends, & significant other. Each item is scored on a scale from 1 to 7 (0 = very strongly disagree, 7 = very strongly agree).
Multidimensional Scale of Perceived Social Support (MSPSS) | Change from Baseline to 3 months
  This scale is a 12-item questionnaire to identify the patients' perceived adequacy of social support from three sources: family, friends, & significant other. Each item is scored on a scale from 1 to 7 (0 = very strongly disagree, 7 = very strongly agree).
Multidimensional Scale of Perceived Social Support (MSPSS) | Change from Baseline to 6 months
  This scale is a 12-item questionnaire to identify the patients' perceived adequacy of social support from three sources: family, friends, & significant other. Each item is scored on a scale from 1 to 7 (0 = very strongly disagree, 7 = very strongly agree).
Multidimensional Scale of Perceived Social Support (MSPSS) | Change from Baseline to 12 months
  This scale is a 12-item questionnaire to identify the patients' perceived adequacy of social support from three sources: family, friends, & significant other. Each item is scored on a scale from 1 to 7 (0 = very strongly disagree, 7 = very strongly agree).
Built Environment | Baseline
  5-items questionnaire to assess the relationship of one's environment to the health outcomes.
Built Environment | Change from Baseline to 3 months
  5-items questionnaire to assess the relationship of one's environment to the health outcomes.
Built Environment | Change from Baseline to 6 months
  5-items questionnaire to assess the relationship of one's environment to the health outcomes.
Built Environment | Change from Baseline to 12 months
  5-items questionnaire to assess the relationship of one's environment to the health outcomes.
Religion/Spirituality | Baseline
  2-items questionnaire to find out the effects of having religion/spiritual beliefs on one's health outcomes.
Religion/Spirituality | Change from Baseline to 3 months
  2-items questionnaire to find out the effects of having religion/spiritual beliefs on one's health outcomes.
Religion/Spirituality | Change from Baseline to 6 months
  2-items questionnaire to find out the effects of having religion/spiritual beliefs on one's health outcomes.
Religion/Spirituality | Change from Baseline to 12 months
  2-items questionnaire to find out the effects of having religion/spiritual beliefs on one's health outcomes.
Oxford Knee Score (OKS) | Baseline
  This 12 items self-reported questionnaire measures patient's pain and level of function. Each item is rated from least to most difficultly or severity. The scoring system ranges from 0 to 4 for each question with 4 representing maximum function and 0 representing poorest function. The lowest (worse) score is 0, and the highest (best) score is 48.
Knee Society Score (KSS) Function | Baseline
  The 3 items patient-reported portion (Function Score) of the KSS covers the patient's mobility (walking distance and stairs) and potential walking aids. Score range of the KSS is from 0 to 100 points for each portion, with higher scores indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Tan, Principal Investigator — Tan Tock Seng Hospital
Locations (3):
- Singapore (3):
  - Khoo Teck Puat Hospital, Singapore
  - St Luke's Eldercare (AMK Polyclinic, Hougang Central, Nee Soon Central), Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Derived] Sahrin R, Ng CJY, Lim CJ, Goh ZZS, Pua YH, Tan BY. Exploring the role of the built environment and psychosocial mediators on knee function in knee osteoarthritis patients in Singapore: a cross-sectional study. BMJ Open. 2024 Nov 2;14(11):e082625. doi: 10.1136/bmjopen-2023-082625. PMID 39488423
- [Derived] Tan BY, Goh ZZS, Lim CJ, Pereira MJ, Yang SY, Tan KG, Tan ACK, Liang P, Abbott JH, Briggs AM, Hunter DJ, Skou ST, Thumboo J, Car J. Singapore KneE osTeoarthritis CoHort (SKETCH): protocol for a multi-centre prospective cohort study. BMC Musculoskelet Disord. 2023 Feb 7;24(1):104. doi: 10.1186/s12891-023-06207-1. PMID 36750930